CLINICAL TRIAL: NCT02591173
Title: Blood Pressure Lowering Effects of Angiotensin-(1-7) in Primary Autonomic Failure
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Difficulty recruiting
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 151461
Record Dates: First submitted 2015-10-27; First posted 2015-10-29 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Autonomic Nervous System Disorders; Pure Autonomic Failure; Shy-Drager Syndrome; Orthostatic Hypotension, Dysautonomic
Keywords: Autonomic; Hypertension; Renin-Angiotensin System
MeSH Terms: conditions — Autonomic Nervous System Diseases; Pure Autonomic Failure; Shy-Drager Syndrome; Hypertension | interventions — angiotensin I (1-7); Acetates; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Angiotensin-(1-7) (Experimental): Patients will receive an intravenous infusion of five ascending doses of Angiotensin-(1-7). The doses are: 1, 2, 4, 8 and 16 ng/kg/min. Each dose will be maintained for 10 minutes, for a total of 50 minutes.
  Interventions: Drug: Angiotensin-(1-7)
- Saline (Placebo Comparator): Patients will receive an intravenous infusion of saline that is matched in volume to the Angiotensin-(1-7) study day. The saline infusion will be maintained for 50 minutes.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Angiotensin-(1-7) — This is a biologically active endogenous angiotensin peptide. It may play an important role in the regulation of blood pressure by dilating blood vessels.
  Other Names: Angiotensin I (1-7); Angiotensin I/II (1-7) Acetate
  Arms: Angiotensin-(1-7)
Drug: Saline — Normal saline will be used as the placebo comparator.
  Other Names: normal saline; 0.9% sodium chloride
  Arms: Saline

SUMMARY:
Pharmacologic approaches to increase levels or actions of the vasodilatory peptide angiotensin-(1-7) are currently in development for the treatment of hypertension based on findings from animal models. There are limited and contradictory clinical studies, however, and it is not clear if this peptide regulates blood pressure in humans. The purpose of this study is to better understand the cardiovascular effects angiotensin-(1-7) in human hypertension, and to examine interactions of this peptide with the autonomic nervous system. The investigators propose that the difficulties in showing angiotensin-(1-7) cardiovascular effects in previous clinical studies relates to the buffering capacity of the baroreceptor reflex to prevent changes in blood pressure. Autonomic failure provides the ideal patient population to test this hypothesis. These patients have loss of baroreflex buffering and have low levels of angiotensin-(1-7) in blood. The investigators will test if angiotensin-(1-7) infusion can lower blood pressure in patients with autonomic failure, and will determine the hemodynamic and hormonal mechanisms involved in this effect.

DETAILED DESCRIPTION:
This is an inpatient study that requires at least four days of admission to the Vanderbilt Clinical Research Center. Autonomic failure patients will be placed on a fixed diet during the admission and will have routine tests performed for screening and clinical characterization. Patients will then receive intravenous angiotensin-(1-7) or saline infusion on two separate study days, with each study day lasting approximately 3 hours. There will be at least one washout day between study days. Patients will be instrumented with two intravenous catheters (one for blood sampling and one for drug infusion), arm and finger blood pressure cuffs, and sticky patches to measure heart rate during the study. The investigators will take baseline measurements of blood pressure and heart rate and collect blood samples. The investigators will also perform a rebreathing test to measure the heart's pumping capacity. After baseline measurements, the investigators will infusion angiotensin-(1-7) or saline for 50 minutes. There will be five doses of angiotensin-(1-7). Each dose will be maintained for 10 minutes. The investigators will measure blood pressure and heart rate, repeat the rebreathing test, and collect blood samples at the end of each dosing period.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of all races between 18 to 80 years of age.
* Diagnosed with primary autonomic failure and supine hypertension. Supine hypertension will be defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 90 mmHg while lying down.
* Able and willing to provide informed consent.

Exclusion Criteria:

* Pregnancy or breast feeding.
* Hemoglobin < 10.5 or hematocrit < 32.
* High-risk patients (e.g. heart failure, symptomatic coronary artery disease, liver impairment, renal failure, history of stroke or myocardial infarction).
* Inability to give or withdraw informed consent.
* Other factors which in the investigator's opinion would prevent the patient from completing the protocol (e.g. clinically significant abnormalities on clinical, mental examination, or laboratory testing or inability to comply with the protocol).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 50 minutes
  The decrease in blood pressure following angiotensin-(1-7) versus saline infusion.

SECONDARY OUTCOMES:
Heart Rate | 50 minutes
  The change in heart rate following angiotensin-(1-7) versus saline infusion.
Cardiac Output | 50 minutes
  The change in cardiac output following angiotensin-(1-7) versus saline infusion.
Stroke Volume | 50 minutes
  The change in stroke volume following angiotensin-(1-7) versus saline infusion.
Systemic Vascular Resistance | 50 minutes
  The change in systemic vascular resistance following angiotensin-(1-7) versus saline infusion.
Renin Activity | 50 minutes
  The change in plasma renin activity following angiotensin-(1-7) versus placebo infusion.
Angiotensin Peptides | 50 minutes
  The change in plasma angiotensin peptides following angiotensin-(1-7) versus placebo infusion.
Aldosterone | 50 minutes
  The change in plasma aldosterone following angiotensin-(1-7) versus placebo infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States